CLINICAL TRIAL: NCT00359944
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Dose-Ranging Study Assessing the Efficacy and Safety of AC-3933 Tablets Twice Daily in Adults With Mild to Moderate Alzheimer's Disease
Brief Title: Safety and Efficacy Study of AC-3933 in Adults With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-3933-271
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 5-(3-methoxyphenyl)-3-(5-methyl-1,2,4-oxadiazol-3-yl)-2-oxo-1,2-dihydro-1,6-naphthyridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AC-3933 (Experimental): AC-3933, 5mg twice daily
  Interventions: Drug: AC-3933
- AC-3933, 20 mg twice daily (Experimental): AC-3933, 20 mg twice daily
  Interventions: Drug: AC-3933
- Placebo (Placebo Comparator): Sugar Pill twice daily
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Drug: AC-3933 — 5mg twice daily
  Arms: AC-3933
Drug: AC-3933 — AC-3933, 20 mg twice daily
  Arms: AC-3933, 20 mg twice daily
Other: Sugar Pill — Sugar Pill twice daily
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate efficacy and safety of different doses of AC-3933 in patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Alzheimer's Disease
* Male or female 55 years or older
* Living with caregiver
* Read, understand and speak English

Exclusion Criteria:

* Need to drive during the study
* Treatment with acetylcholinesterase inhibitors or NMDA antagonist, such as Aricept or Namenda, within 2 weeks of check-up and during the study
* Frequent Smoker
* Frequent Consumer of Caffeine

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (34):
- United States (34):
  - Clinical Trials Inc., LIttle Rock, Alaska
  - PsyPharma Clinical Research Inc., Phoenix, Arizona
  - ClinicalStudies Center LLC, Little Rock, Arkansas
  - Vertex Clinical Research, Bakersfield, California
  - East Bay Physicians Medical Grou[, Berkeley, California
  - Margolin Brain Institute, Fresno, California
  - Clinical Trials Associates, Mission Viejo, California
  - University of California, Orange, California
  - Pacific Research Network, San Diego, California
  - Memory Disorder Clinic, Deerfield Beach, Florida
  - Berma Research Group, Hialeah, Florida
  - Advanced Research Institute of Miami, Miami, Florida
  - Research Institute of Miami, Miami, Florida
  - Research Center of Florida Inc., Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Compass Research LLC, Orlando, Florida
  - Department of Psychiatry and Behavioral Medicine, Tampa, Florida
  - Stedman Clinical Trials LLC, Tampa, Florida
  - Four Rivers Clinical Research Inc., Paducah, Kentucky
  - Northern Michigan Neurology, Traverse City, Michigan
  - Minneapolis, Minnesota
  - Clinical Psychopharmacology Consultants PA, Saint Louis Park, Minnesota
  - Precise Research Centers INc., Flowood, Mississippi
  - Psych Care Consultants Research, St Louis, Missouri
  - Odyssey Researcfh, Fargo, North Dakota
  - Paradigm Research Professionals LLP, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - UT Medical Group Inc., Memphis, Tennessee
  - Neurological Research Center, Inc., Bennington, Vermont
  - International Clinical Research Associates LLC, Richmond, Virginia
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
  - Internal Medicine Northwest, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 patients were excluded from analysis because of QA issues at a study site.
Groups:
- AC-3933, 5 mg: AC-3933, 5mg twice daily
- AC-3933, 20 mg: AC-3933, 20 mg twice daily
Period: Overall Study
Arm/Group | AC-3933, 5 mg | AC-3933, 20 mg | Placebo
Started | 50 | 47 | 57
Completed | 34 | 28 | 38
Not Completed | 16 | 19 | 19

BASELINE CHARACTERISTICS:
Population: 132 subjects were from the full analysis set, which was defined as all randomized subjects who took at least one dose of study drug and had greater than/equal to one post-baseline ADAS-Cog assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-3933 | AC-3933, 20 mg | Placebo | Total
Number analyzed (Participants) | 43 | 40 | 49 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 43 | 40 | 49 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 75.5 (8.57) | 74.8 (9.54) | 76.3 (8.73) | 75.6 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 38 | 95
  Male | 13 | 13 | 11 | 37
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 49 | 132

OUTCOME MEASURES:

1. Primary Outcome: Total Score of Alzheimer's Disease Assessment Scale - Cognition Subscale (ADAS-COG)From Best Total Score (0) to Worst Total Score (70)
Description: Change from baseline to week 16 of the double blind treatment in the Alzheimer's Disease Assessment Scale - Cognition Subscale (ADAS-COG) total score The Alzheimer's Disease Assessment Scale if used for assessing the severity of dysfuncion and for research in patients with AD, particularly in clinical drug trials. It consists of 11 items testing orientatin, memory, word usage and recognition, receptive speech, spatial abilities, ideational praxis, ability to follow instructions, spontanious speech abilities, and comprehension. The higher the overall score (maximum 70), the more severe the dysfunction/impairment.
Time Frame: Baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-3933, 5 mg | AC-3933, 20 mg | Placebo
Number analyzed (Participants) | 43 | 40 | 49
units on a scale | -1.3 (0.84) | -2.9 (0.88) | -1.5 (0.78)

2. Secondary Outcome: Clinicians Interview Based Impression of Change (CIBIC)-Plus
Description: Clinicians Interview Based Impression of Change (CIBIC)-Plus-Plus scores at week 16 of the double blind treatment.
  CIBIC-Plus is ranged between 1 and 7 (1=very much improved, 4=no change, and 7=very much worsened). We were expecting smaller value of CIBIC-Plus at the study end.
Time Frame: Baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-3933, 5 mg | AC-3933, 20 mg | Placebo
Number analyzed (Participants) | 43 | 40 | 49
units on a scale | 4.1 (0.97) | 3.9 (1.11) | 3.9 (0.91)

3. Secondary Outcome: Disability Assessment for Dementia (DAD)
Description: Change from baseline to week 16 of the double blind treatment in the Disability Assessment for Dementia (DAD) scores.
  The DAD is administered as a clinician-assisted interview with the caregiver and was developed to assess functional abilities in ADLs in community-dwelling dementia patients. The scale consists of 40 questions assessing basic and instumental ADLs. A total score is obtained by adding the rating for each question and converting this total score out of 100. The items rated N/A are not considered for the total score. Higher scores represent less disability in activities of daily living (ADL) while lower scores indicate more dysfunction.
Time Frame: Baseline to 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-3933, 5 mg | AC-3933, 20 mg | Placebo
Number analyzed (Participants) | 43 | 40 | 49
units on a scale | -2.7 (1.89) | 4.0 (2.10) | 4.2 (1.80)

ADVERSE EVENTS:
Time Frame: February 2006 to September 2008
Description: The AE summary was based on the safety population, which was defined as all randomized patients who received at least one dose of the study drug (58 placebo, 50 AC-3933 5mg, 46 AC-3933 20mg. Once subject randomized to AC-3933 20mg group received placebo during the course of the study. So this subject was summarized in the placebe group.
Arm/Group | AC-3933, 5 mg | AC-3933, 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/50 | 4/46 | 5/58
Other Adverse Events (participants affected / at risk) | 11/50 | 12/46 | 17/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-3933, 5 mg (N=50) | AC-3933, 20 mg (N=46) | Placebo (N=58)
Cardiac Failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Colon Cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Abnormal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-3933, 5 mg (N=50) | AC-3933, 20 mg (N=46) | Placebo (N=58)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5)
Urinary Tract infection (Infections and infestations) | 2 (2) | 2 (2) | 5 (5)
Electroencephalogram abnormal (Investigations) | 1 (1) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No